CLINICAL TRIAL: NCT05888272
Title: Examining the Effect of Stress Management Training on the Business Performance of Women Entrepreneurs in Ethiopia
Brief Title: Addressing Stress Among Women Entrepreneurs in Ethiopia - Scale up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: World Bank (Other)
Collaborators: Ethiopian Medical Association (Unknown); Policy Studies Institute (Unknown); Addis Ababa University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DWMTS-Scaleup
Record Dates: First submitted 2023-04-15; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Mental Stress; Stress; Stress, Job; Emotion Regulation; Violence, Gender-Based; Economic Problems
Keywords: Stress Managment; Psychological Wellbeing; Business Performance; Intimate Partner Violence
MeSH Terms: conditions — Stress, Psychological; Occupational Stress; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Study participants that meet the eligibility criteria are randomly assigned to the intervention and waitlist control groups.
Who Masked: Outcomes Assessor
Masking Description: Randomized using computer-generated randomization at one point in time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Stress Managment (Experimental): A locally adapted self-help guidebook originally developed by the World Health Organization (WHO), 'Doing what matters in times of stress' for managing disruptive emotions and psychological distress, will be delivered to women entrepreneurs at their residences, followed by 7 phone calls from a trained mental health helper to reinforce the materials over a 10-week period. The intervention is intended to help people manage their psychological distress associated with a range of adversities but is not intended for participants with severe mental health problems such as psychosis or imminent risk of suicide
  Interventions: Behavioral: Stress managment
- Waitlist Control (No Intervention): This group will receive the DWMTS handbook if the study documents a positive impact on the outcomes of interest.

INTERVENTIONS:
Behavioral: Stress managment — The Doing What Matters in Times of Stress self-help manual materials and lay helper scripts utilized in the study are rooted in the principles of Acceptance and Commitment Therapy (ACT). They are designed to improve psychological flexibility which refers to an individual's ability to adapt to changing situations, reallocate mental resources, shift perspectives, and balance competing priorities. The ACT approach teaches individuals how to manage challenging thoughts and emotions through mindfulness techniques, while also guiding them to live in alignment with their personal values.
  Other Names: Doing What Matters in Times of Stress self-help hand book - the intervention does not involve any drugs.
  Arms: Experimental - Stress Managment

SUMMARY:
The objective of this study is to examine the impact of the "Doing What Matters in Times of Stress" guided self-help handbook, along with phone-based lay helpers sessions, on the psychological well-being, business performance, and incidence of intimate partner violence among women entrepreneurs in Ethiopia.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of the "Doing What Matters in Times of Stress Guided" self-help manual on mental distress, business performance, and intimate partner violence experienced by women entrepreneurs in Ethiopia. The study will be conducted in four cities - Addis Ababa, Hawassa, Bahir Dar, and Adama - using a randomized controlled trial (RCT) design. The investigators will screen 5000 potential participants via phone and enroll 1200 eligible women, who will be equally distributed across the four cities. After an in-person baseline survey, the women will be stratified by marital status and city and randomized into the intervention or waitlist control group using a computer-generated random assignment. The intervention group will receive seven phone-based sessions over ten weeks to review the self-help manual materials with a lay helper. Two follow-up surveys will be conducted after the intervention, the first one a month after the completion of the intervention, and the second one twelve months after completion.

This study is a continuation of a pilot study conducted between July 2021 and August 2022 (PRS registration ID - NCT05208723). The current study seeks to build on the pilot study in the following dimensions:

1. Increase the sample size to 1200 women entrepreneurs to improve the power of the study to detect the impact of the intervention on business performance outcomes,
2. Widen the geographical and contextual coverage,
3. Allow entrepreneurs to invite a household member to attend the self-help phone sessions with them,
4. Capture the impact on intimate partner violence,
5. Introduce a short conflict module to capture the direct and indirect effects of conflict on mental health outcomes, business performance, and intimate partner violence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18;
* Those who plan to live in the study city in the next six months;
* Those who can read and speak Amharic and can understand the study questionnaire;
* Those who have the capacity to provide informed consent;
* Score 8 or above on the Ethiopian adaptation of Kessler-6

Exclusion Criteria:

* Kessler 6 score >20;
* Those who have recent or current suicidal thoughts or plans;
* Those who have limitations in understanding the study questionnaire;
* Those who do not have the capacity to provide informed consent;
* Do not have access to a phone;
* Not interested in receiving the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifying as women
Enrollment: 1200 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mental Distress using the Kessler Psychological Distress Scale (K-6) | Time Frame: 4-6 weeks post intervention
  Minimum value of 0 and a maximum value of 24. Higher scores indicate high levels of psychological distress (worse outcome)
Mental Distress using the Kessler Psychological Distress Scale (K-6) | Time Frame:12 months post intervention
  Minimum value of 0 and a maximum value of 24. Higher scores indicate high levels of psychological distress (worse outcome)
Depression using the Patient Health Questionnaire (PHQ-9) | Time Frame: 4-6 weeks post intervention
  Minimum score 0 and a maximum score of 27. Higher scores indicate increased levels of depressive symptoms (worse outcome).
Depression using the Patient Health Questionnaire (PHQ-9) | Time Frame: 12 months post intervention
  Minimum score 0 and a maximum score of 27. Higher scores indicate increased levels of depressive symptoms (worse outcome).
Stress using the Perceived Stress Scale | Time Frame: 4-6 weeks post intervention
  Minimum score of 0 and a maximum of 40. Higher scores indicate high levels of perceived stress (worse outcome). Investigators will reverse code items 4,5, 7 and 8
Stress using the Perceived Stress Scale | Time Frame: 12 months post intervention
  Minimum score of 0 and a maximum of 40. Higher scores indicate high levels of perceived stress (worse outcome). Investigators will reverse code items 4,5, 7 and 8
Self-Esteem using the Rosenberg Self-esteem Scale | Time Frame: 4-6 weeks post intervention
  Minimum score 10 and a maximum score of 40. Investigators will reverse code items 3,5,8,9 and 10 . Higher scores indicate high levels of self-esteem (better outcome)
Self-Esteem using the Rosenberg Self-esteem Scale | Time Frame:12 months post intervention
  Minimum score 10 and a maximum score of 40. Investigators will reverse code items 3,5,8,9 and 10 . Higher scores indicate high levels of self-esteem (better outcome)
World Health Organisation- Five Well-Being Index (WHO-5) | Time Frame: 4-6 weeks post intervention
  Minimum score of 0 and a maximum of 25. Higher scores mean better wellbeing (better outcome). Scores are transformed to 0-100 (by multiplying by 4.
World Health Organisation- Five Well-Being Index (WHO-5) | Time Frame: 12 months post intervention
  Minimum score of 0 and a maximum of 25. Higher scores mean better wellbeing (better outcome). Scores are transformed to 0-100 (by multiplying by 4.
Functional Impairment using the World Health Organization Disability Assessment Schedule (WHODAS-2.0 -12 item version) | Time Frame: 4-6 weeks post intervention
  Minimum score of 12 and a maximum of 60. Higher scores indicate high levels of disability (worse outcome)
Functional Impairment using the World Health Organization Disability Assessment Schedule (WHODAS-2.0 -12 item version) | Time Frame: 12 months post intervention
  Minimum score of 12 and a maximum of 60. Higher scores indicate high levels of disability (worse outcome)

SECONDARY OUTCOMES:
Business Performance 1 | Time Frame: 12 months post intervention
  Monthly Profits
Business Performance 2 | Time Frame: 12 months post intervention
  Monthly Sales
Business Performance 3 | Time Frame: 12 months post intervention
  Business size measured using number of employees
Intimate Partner Violence 1 | Time Frame: 12 months post intervention
  Experience of at least one form of Physical Violence measured using the Demographic and Health Survey module for the experience of physical intimate partner violence.
Intimate Partner Violence 2 | Time Frame: 12 months post intervention
  Experience of at least one form of Emotional Violence measured using the Demographic and Health Survey module for the experience of emotional intimate partner violence.

CONTACTS AND LOCATIONS:
Overall Officials: Adiam Hagos Hailemicheal, MSc, Principal Investigator — World Bank; Naira Kalra, PhD, Principal Investigator — World Bank; Medhin Selamu Tegegn, PhD, Principal Investigator — Addis Ababa University; Kassahun Habtamu Mekonnen, PhD, Principal Investigator — Addis Ababa University
Locations (1):
- Policy Studies Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified IPD two years after the completion of each survey based after securing clearance from the Ethiopian Public Health Asssociations IRB.
Time Frame: Baseline survey - April, 2025; Follow up surveys - July, 2025
Access Criteria: The data will be publicly available on the World Bank's microdata website. Use of the dataset must be acknowledged using a citation which would include:
  1. the identification of the Principal Investigators,
  2. the title of the survey (including country, acronym and year of implementation)
  3. the survey reference number
  4. the source and date of download
URL: https://www.worldbank.org/en/programs/africa-gender-innovation-lab/brief/africa-gender-innovation-lab-data